CLINICAL TRIAL: NCT02605759
Title: Clinical Study to Evaluate the Safety, Feasibility and Efficacy of the Coldplay CryoBalloon Focal Ablation System for the Cryoablation of Dysplastic Squamous Tissue in Patients With Esophageal Squamous Cell Dysplasia
Brief Title: Coldplay Cryoablation of Dysplastic Squamous Tissue in Patients With Esophageal Squamous Cell Dysplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pentax Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-0013
Record Dates: First submitted 2015-11-13; First posted 2015-11-16 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Esophageal Squamous Cell Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CryoBalloon Focal Ablation System (Experimental): CryoBalloon Focal Ablation for the treatment of esophageal squamous cell dysplasia
  Interventions: Device: CryoBalloon Focal Ablation System

INTERVENTIONS:
Device: CryoBalloon Focal Ablation System — Positioned within the esophagus at the target location, the Balloon is simultaneously inflated and cooled with nitrous oxide. The nitrous oxide cools the inner Balloon surface. The Balloon remains stationary during the delivery of the nitrous oxide for the Cryoablation of Dysplastic Squamous Tissue in Patients with Esophageal Squamous Cell Dysplasia
  Other Names: C2 CryoBalloon Focal Ablation System; Coldplay CryoBalloon Focal Ablation System

SUMMARY:
To demonstrate the feasibility, safety and efficacy of the CryoBalloon Ablation System for the treatment of esophageal squamous cell dysplasia.

DETAILED DESCRIPTION:
Multi-center, prospective, single arm, non-randomized study. The study will proceed in two phases: a pilot phase, followed by the feasibility, safety and efficacy phase. In the pilot phase, up to five (5) patients at one (1) site will be treated with the CryoBalloon Ablation System to confirm its safety and feasibility in the treatment of squamous dysplasia. The second phase will be conducted at two (2) centers and will enroll up to 50 subjects to evaluate the feasibility, safety and efficacy of the CryoBalloon Ablation System for the treatment of squamous dysplasia.

ELIGIBILITY:
Inclusion Criteria:

* At least one unstained lesion (USL) in the esophagus upon high resolution endoscopy with Lugol's staining
* Flat (type 0-IIb) appearance of the USL
* Total area of USLs is a maximum longitudinal size of 6cm and covering a maximum of one-half of the circumference of the esophagus
* Proven (by histopathological analysis) medium-grade or high-grade intraepithelial neoplasia (MGIN or HGIN) in at least one USL
* Older than 18 years of age at time of consent
* Operable per institution's standards
* Provides written informed consent on the Ethics Committee-approved informed consent form
* Willing and able to comply with study requirements for follow-up

Exclusion Criteria:

* Esophageal stenosis or stricture preventing advancement of a therapeutic endoscope within 4cm of the treatment zone
* Other USLs containing MGIN, HGIN, or ESSC outside the designated treatment area
* Any previous ablative therapy in the esophagus (photodynamic therapy, multipolar electrical coagulation, argon plasma coagulation, laser treatment) or any radiation therapy to the esophagus
* Any previous esophageal surgery (except anti-reflux surgery)
* Any cancer (squamous cell or non-squamous cell) within the previous five (5) years
* Active inflammation in the treatment zone due to esophageal reflux, as confirmed by endoscopic examination
* Known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent, post-treatment instructions or follow-up guidelines
* Pregnant or planning to become pregnant during the study follow-up period
* Life expectancy ≤2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03; Primary Completion 2018-01-27 (Actual); Study Completion 2018-01-27 (Actual)

PRIMARY OUTCOMES:
Serious, device-related adverse events | Day 30
  Incidence of serious, device-related adverse events
Successful, complete ablation of the unstained lesions (USLs) within the treatment area (TA) | Day 0
  The percentage of subjects with successful, complete ablation of the USLs within the TA as determined by the endoscopist at the time of the treatment endoscopy(s)
Percentage of subjects with absence of ULS containing medium-grade intraepithelial neoplasia (MGIN) or high-grade intraepithelial neoplasia (HGIN) within the original TA | 3 months
  Percentage of subjects with absence of ULS containing medium-grade intraepithelial neoplasia (MGIN) or high-grade intraepithelial neoplasia (HGIN) within the original TA at three (3) months following endoscopic cryoablation. This will be evaluated by visual endoscopic exam and two (2) biopsies negative for squamous epithelial dysplasia confirmed by histopathological analysis

SECONDARY OUTCOMES:
Absence of USLs containing MGIN, HGIN or cancer | 12 months
  Efficacy defined as the absence of USLs containing MGIN, HGIN or cancer within the original TA after the last endoscopic ablation.
Complete eradication after one treatment | 12 months
  Percentage of subjects achieving complete eradication after one treatment session with the CryoBalloon Ablation System
Device performance | Day 0
  Device performance, assessed by Device malfunction
Procedure time | Day 0
  Procedure time, defined as the time from the introduction of the endoscope to its removal
Adverse Events | 12 Months
  Incidence of all treatment-related and serious, non-device related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Guiqi Wang, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ke Y, van Munster SN, Xue L, He S, Zhang Y, Dou L, Liu Y, Liu X, Liu Y, Li W, Lv N, Dawsey SM, Weusten BLAM, Bergman JJGHM, Wang G. Prospective study of endoscopic focal cryoballoon ablation for esophageal squamous cell neoplasia in China. Gastrointest Endosc. 2019 Aug;90(2):204-212. doi: 10.1016/j.gie.2019.03.017. Epub 2019 Mar 25. PMID 30922862